CLINICAL TRIAL: NCT07073196
Title: Single Implant Crowns Supported by Narrow or Standard Diameter Implants in Molar Sites: a Randomized Controlled Trial
Brief Title: Single Implant Crowns Supported by Narrow or Standard Diameter Implants in Molar Sites
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed Bin Rashid University of Medicine and Health Sciences (Other)
Responsible Party: Principal Investigator, Momen Atieh, Professor, Mohammed Bin Rashid University of Medicine and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MBRUMHS - June 2025; MBRU IRB-2025-110 (Other: MBRU)
Record Dates: First submitted 2025-06-28; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Dental Implants
Keywords: Dental implants

STUDY DESIGN:
Intervention Model Description: Prospective, in which participants will be recruited and then followed up throughout a specified period of time.
  Randomized, parallel designed, concurrent controlled trial with participants randomly allocated to either test or control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narrow implants (Experimental): Narrow implants diameter 3.3 mm to replace missing molar tooth
  Interventions: Procedure: Dental implant treatment (narrow implants)
- Standard implants (Active Comparator): Standard implants diameter 4.5 mm to replace missing molar tooth
  Interventions: Procedure: Dental implant treatment (standard implants)

INTERVENTIONS:
Procedure: Dental implant treatment (narrow implants) — Replacement of a missing molar tooth with a narrow dental implant
  Arms: Narrow implants
Procedure: Dental implant treatment (standard implants) — Replacement of a missing molar tooth with a standard dental implant
  Arms: Standard implants

SUMMARY:
Standard dental implants require sufficient bone and spacing, which may not be available in all patients. To address these limitations, narrow diameter implants (≤3.5 mm) have been introduced as a less invasive alternative, especially useful for medically compromised patients or those avoiding bone grafts. However, narrow implants made of pure titanium have shown long-term biological and technical concerns.

The introduction of titanium-zirconium (TiZr) alloy has improved mechanical strength, and several studies have demonstrated favorable outcomes with narrow TiZr implants. Yet, evidence remains limited regarding their exclusive use in high-load posterior (molar) regions. Prior studies report conflicting failure rates, potentially linked to prosthetic design and occlusal forces, but lack quantitative analysis of bite forces or prosthetic angles.

Emergence angle, prosthetic platform width, and implant-abutment connection may all influence implant stability and peri-implant tissue health. A newly introduced TorcFit™ connection may offer better stress distribution and torque resistance, but its clinical relevance-especially in narrow implants used for molars-remains untested.

DETAILED DESCRIPTION:
Introduction (background and research question)

Standard diameter dental implants require sufficient bone volume and adequate interdental distance to prevent adverse bone level changes, or unfavorable long-term esthetic outcomes. To overcome site specific limitations, simplify treatment protocols, and expand clinical applications, short (< 10 mm) and narrow diameter (≤ 3.5 mm) implants were introduced. It has been suggested that narrow diameter dental implants would allow a less invasive surgical procedure by reducing the need for bone augmentation, a viable option for medically compromised patients and those averse to the use of bone grafting materials. However, the use of narrow diameter implants of commercially pure titanium (cpTi) has been associated with several biological and technical concerns when used over a long period of function.

The use of titanium and zirconium (TiZr) alloy improved the mechanical properties and several clinical studies showed that narrow diameter TiZr implants had high survival rates and comparable performance to standard diameter cpTi implants across various clinical indications. The clinical outcomes of narrow diameter TiZr were also comparable to standard diameter implants of the same TiZr material when replacing single missing teeth in the anterior or posterior regions of the maxilla or mandible. On the other hand, the use of narrow diameter TiZr implants to support single crown restorations exclusively in the posterior region remains limited. One randomized controlled trial has reported on the clinical outcomes of single narrow (3.3 mm) diameter TiZr implants in molar sites. These studies reported failure rates of 1% and 18% at one- and three-year follow-up, respectively. The failed narrow diameter implants were regular neck (RN) with prosthetic platform of 4.8 mm and were mostly lost because of implant fracture below the internal screw channel. Traumatic occlusal forces were thought to be the reason behind these failures. However, the occlusal wear or the bite forces on these narrow implant-supported crowns were not quantitatively assessed.

While it could be speculated that the wider prosthetic platform of 4.8 mm diameter might have caused unfavorable leverage on the narrow diameter implant body placed in sites of high occlusal load (i.e., single molar sites), wider prosthetic platform in molar sites may provide favorable prosthetic design and emergence profile that could be associated with greater stability of peri-implant hard and soft tissues. Different prosthetic-related factors, particularly the restorative angles and emergence profile, may have significant impact on marginal mucosal and bone levels and increase the risk of developing peri-implantitis. Narrow diameter implants might be associated with implant restorations with an emergence angle of > 30° in molar sites. The long-term outcomes of implant restorations with different emergence angles were recently evaluated in a systematic review. While significant differences were not observed in terms of periodontal and esthetic outcomes, the authors concluded that platform-matched implant restorations with an emergence angle of ≤ 30° might be associated with less changes in peri-implant marginal bone levels when compared to implant restorations with an emergence angle of > 30°. However, the evidence support was of low to moderate certainty and further studies are still required.

Another reason that has been implicated in the biological and technical complications of dental implants is the poor fit and instability of the implant-abutment connection. Narrow diameter Straumann tissue level dental implants have 15° internal cone with either four internal CrossFit® grooves or 8° morse taper synOcta® connection. These configurations allow flexible positioning of the prosthetic components but evidence on using narrow diameter implants with either CrossFit® or synOcta® connection in molar sites remains insufficient. Recently, a new implant-abutment connection has been introduced with the premise of ensuring transmission of high torques. The stability of the new TorcFit™️ implant-abutment connection was shown to be similar to that of the CrossFit® connection. However, the TorcFit™️ connection, with its 7° conical connection and six-sided star-shaped anti-rotational element, may allow transmission of higher torques, maintain a flexible alignment of the prosthetic components, and ensure uniform stress distribution. It is yet to seen to what extent this new implant-abutment connection influences the clinical performance of a narrow (3.3 mm) or standard (4.5 mm) diameter implant in the replacement of single missing molars.

Aim(s) of the study:

The objectives of this single-center three-year randomized controlled trial will be:

To evaluate the clinical, and radiographic outcomes of narrow and standard diameter TiZr implants used to support screw-retained monolithic zirconia crowns in molar sites.

To evaluate the long-term effects of the restorative emergence angle on the peri-implant mucosal level, marginal bone level, periodontal parameters and prevalence of biological complications.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years.
* Require replacement of single missing molar tooth with dental implant in fully healed sites.
* Controlled oral hygiene (full-mouth plaque and bleeding scores ≤ 25% at baseline).
* Intact adjacent teeth and opposing dentition.
* Fully healed sites (≥ 6 months) with limited bone availability in the horizontal bucco-lingual dimension (residual bone width of ≤ 6 mm) and minimal height of 8 mm.
* Good compliance and commitment to attend follow-up review appointments.
* Willing to provide informed consent.

Exclusion Criteria:

* Localized/generalized periodontitis.
* Any medical condition that may contraindicate implant treatment (Bornstein et al., 2009).
* Bone metabolic disease and/or taking medications that affect bone metabolism.
* Long term use of non-steroidal anti-inflammatory medications.
* History of malignancy, radiotherapy or chemotherapy.
* Pregnant or lactating women.
* Smokers.
* Severe bruxism or parafunctional habits.
* Large occlusal discrepancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Peri-implant mucosal recession rate | Peri-implant mucosal recession rate will be assessed at three and twelve months
  The peri-implant mucosal margin will be assessed by measuring the clinical crown height and recorded as yes/no

SECONDARY OUTCOMES:
Emergence angle of implant restorations | Three months
  Emergence angle of implant restorations will be measured on radiographs by recording the angle between the implant long axis and a line tangent to implant restorations
Implant success/survival rate | After 12 months and annually for three years
  Implant success/survival rate will be assessed clinically after one year of implant restoration and annually up to three years. A successful implant is the one that will meet the criteria proposed by the European Federation of Periodontology (Albrektsson and Isidor, 1994), while a survived implant is the one that will remain in function but without meeting the success criteria. An implant is considered failed when it will be removed.
Changes in peri-implant marginal bone level | Three and twelve months
  Changes in peri-implant marginal bone level will be assessed standardized periapical radiographs.
Implant stability measurements | Baseline, three and twelve months
  Implant stability measurements will be recorded using an electronic handheld device (Osstell Beacon, W&H, Göteborg, Sweden). The device uses the resonance frequency analysis (RFA) to measure the implant stiffness in implant stability quotient (ISQ) units (Sennerby and Meredith, 1998, Sennerby and Meredith, 2008). The ISQ scale ranges from 0 to 100 with values higher than 65 ISQ indicating a satisfactory implant stability (Atieh et al., 2012, Atieh et al., 2014, Sennerby and Meredith, 2008).
Need for bone augmentation | Baseline
  Need for bone augmentation with autogenous bone chips, xenograft and resorbable collagen membrane, as described by Buser and co-workers (2009) recorded as yes/no.
The width and height of keratinized tissue | At three months of implant restoration and then annually up to three years.
  The width and height of keratinized tissue (Lang and Berglundh, 2011) will recorded using a manual periodontal probe (UNC-15 periodontal probe, Hu-Friedy®, Chicago, USA) and endodontic file (ISO 15).
Prosthetic outcome | At 12 months and annually for three years.
  Prosthetic outcome will be determined using a modified United States Public Health Service (USPHS) criteria (Bayne and Schmalz, 2005, Muhlemann et al., 2020). Each crown will be assessed on 12 parameters: patient satisfaction, ceramic fracture/chipping, abutment screw loosening, abutment screw fracture, debonding of titanium base abutment, fracture of titanium base abutment, loss of screw access restoration, marginal fit of abutment to implant, proximal contacts, occlusal contact, color match to neighboring teeth/restorations and opposing tooth/restoration fracture.

CONTACTS AND LOCATIONS:
Locations (1):
- MBRU, Dubai, United Arab Emirates